CLINICAL TRIAL: NCT01677988
Title: Phase II Study of Neoadjuvant Folfirinox Chemotherapy Followed by Capecitabine With Concurrent Limited Field Radiation Therapy in Patients With Localized Pancreatic Head Adenocarcinoma
Brief Title: Neoadjuvant Folfirinox Followed by Capecitabine and Limited Field Radiation for Localized Pancreatic Head Adenocarcinoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was terminated due to low accrual.
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Principal Investigator, Paul O'Brien, Assistant Professor, Medical University of South Carolina
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 101822
Record Dates: First submitted 2012-08-29; First posted 2012-09-03 (Estimated); Results first posted 2016-01-15 (Estimated); Last update posted 2016-01-15 (Estimated); Status verified 2015-07

CONDITIONS: Adenocarcinoma of Head of Pancreas
Keywords: NEOADJUVANT FOLFIRINOX CHEMOTHERAPY; LOCALIZED PANCREATIC HEAD ADENOCARCINOMA; RADIATION THERAPY
MeSH Terms: interventions — Chemoradiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Chemotherapy, Chemoradiation, Surgery (Experimental): Neoadjuvant Chemotherapy- Modified FOLFIRINOX chemotherapy Day 1 and Day 15 of 28 day cycles for 3 cycles with growth factor support Chemoradiation Surgical Resection
  Interventions: Drug: Neo-adjuvant Chemotherapy; Radiation: Chemoradiation; Procedure: Surgical Resection

INTERVENTIONS:
Drug: Neo-adjuvant Chemotherapy — 1. Modified FOLFIRINOX chemotherapy Day 1 and Day 15 of 28 day cycles, for three (3) cycles with growth factor support.
  2. Restaging # 1. (CT or MRI; use same modality as baseline staging unless otherwise indicated by Study Team)
     1. Progressive Disease (PD) → Off study. Subsequent treatment per patient's primary MD.
     2. Stable Disease (SD) or Tumor Response → Continue to Registration #2 for Chemoradiation.
  Other Names: FOLFIRINOX chemotherapy
Radiation: Chemoradiation — 1. Chemoradiation may be administered at selected approved CTN sites.
  2. Determination of resectability as reviewed and documented by MUSC-HCC GI Tumor Board.
     1. Unresectable → Off study. Subsequent treatment per patient's primary MD.
     2. Resectable → Continue to Registration #3 for Surgical Resection
Procedure: Surgical Resection — 1. Meets criteria for resectable* →pancreaticoduodenectomy (POD)
  2. At time of resection, snap frozen tumor specimen sent for correlative biomarker studies

SUMMARY:
This study is for subjects with adenocarcinoma of the pancreas. The purpose of this research study is to determine the safety and effectiveness of modified Folfirinox and radiation therapy as treatment for adenocarcinoma (cancer) of the pancreas before surgery. Screening tests will be done to determine if subjects are eligible for participation in this study. If subjects are eligible to participate and agree to participate they will begin chemotherapy. After 3 cycles of chemotherapy, subjects will begin chemoradiation. Within 4 to 8 weeks of completing radiation therapy, subjects will have surgery. There will also be post-treatment and follow-up evaluations. Subjects will be followed for every 3 months for 3 years after their initial registration.

ELIGIBILITY:
Inclusion Criteria:

* Patient has histologically or cytologically confirmed borderline resectable adenocarcinoma of the pancreas. Patients with islet cell or other neuroendocrine neoplasms are excluded.
* Borderline resectable disease as outlined in the protocol
* ≥ 18 years of age.
* Male or non-pregnant and non-lactating female. If a female patient is of childbearing potential, she must have a negative serum pregnancy test (β hCG) documented within 72 hours of the first administration of study drug.
* If sexually active, the patient must agree to use contraception considered adequate and appropriate by the Investigator.
* Patient must not have received prior chemotherapy or radiation for pancreatic cancer and no exposure to systemic chemotherapy.
* Patient have acceptable blood counts, chemistries & coagulation at baseline as outlined in the protocol
* Patient has an ECOG performance status PS 0-1.
* Patient has been informed about the nature of the study and has agreed to participate in the study and signed the Informed Consent Form prior to participation in any study-related activities.
* Endoscopic ultrasound (EUS) with FNA for cytology.
* Patients should not have any evidence of active or uncontrolled infection requiring treatment with antibiotics.

Exclusion Criteria:

* Patient has localized resectable, locally advanced unresectable or advanced metastatic disease. Patients with adenocarcinoma of the pancreatic body or tail are ineligible.
* Patient has active, uncontrolled bacterial, viral, or fungal infection(s) requiring systemic therapy.
* Patient has known infection with HIV.
* Patient has undergone major surgery, other than diagnostic surgery (i.e.surgery done to obtain a biopsy for diagnosis without removal of an organ), within 4 weeks prior to Day 1 of treatment in this study.
* Prior chemotherapy, immunotherapy or radiation for pancreatic cancer.
* Patient has a history of allergy or hypersensitivity to the study drugs.
* Patient has serious medical risk factors involving any of the major organ systems such that the Investigator considers it unsafe for the patient to receive chemotherapy and/or radiation therapy.
* Patients must not require chronic use of immunosuppressive agents (e.g. methotrexate, cyclosporine).
* No other prior malignancy is allowed except for the following: adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, adequately treated Stage I or II cancer from which the patient is currently in complete remission, or any other cancer from which the patient has been disease-free for five years.
* Patients must not have clinically significant cardiovascular disease (including myocardial infarction, unstable angina, symptomatic congestive heart failure, serious uncontrolled cardiac arrhythmia) < 1 year before randomization.
* Patients must not have a history of any medical or psychiatric condition or laboratory abnormality that in the opinion of the investigator may increase the risks associated with the study participation or investigational product(s) administration or may interfere with the interpretation of the results.
* Patient is unwilling or unable to comply with study procedures.
* Patient is enrolled in any other therapeutic clinical protocol or investigational trial.
* Patients aged > 70

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2012-07; Primary Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul E. O'Brien, MD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Chemotherapy, Chemoradiation, Surgery: Neoadjuvant chemotherapy - modified FOLFIRINOX chemotherapy Day and and Day 15 of 28 days cycles for 3 cycles with growth factor support followed by chemoradiation for 6-8 weeks, then surgical resection
Period: Overall Study
Arm/Group | Chemotherapy, Chemoradiation, Surgery
Started | 3
Completed | 1
Not Completed | 2
Not completed — Lack of Efficacy | 2

BASELINE CHARACTERISTICS:
Arm/Group | Chemotherapy, Chemoradiation, Surgery
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 3
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Estimate the R0/R1 Resection Rate
Description: Estimate the R0/R1 resection rate as the proportion of patients with R0 or R1 resection status based on the ITT population. R0 resection status is macroscopic complete removal of tumor by non-contaminated operation, with neither macroscopic nor microscopic residual tumor. R1 resection status is macroscopic complete removal of tumor by non-contaminated operation, with microscopic residual tumor.
Time Frame: at time of surgery
Population: Only subjects who had surgery were included in the outcome measure data.
Measure: Number; unit: participants
Groups:
- Chemotherapy, Chemoradiation, Surgery: Neoadjuvant chemotherapy - modified FOLFIRINOX chemotherapy Day and and Day 15 of 28 days cycles for 3 cycles with growth factor support followed by chemoradiation for -08 weeks, then surgical resection
Arm/Group | Chemotherapy, Chemoradiation, Surgery
Number analyzed (Participants) | 1
participants
  R0 resection status | 1
  R1 resection status | 0

2. Secondary Outcome: Radiographic Tumor Response
Description: The rate of CR, PR, SD and PD will be estimated as described in Section 14B prior to chemoradiation start and prior to surgery. The analysis population for estimation of radiographic response rate will be the ITT population.
Time Frame: From enrollment to Surgery
Population: All subjects enrolled and had a response assessment are included in the outcome measure below.
Measure: Number; unit: participants
Arm/Group | Chemotherapy, Chemoradiation, Surgery
Number analyzed (Participants) | 3
participants
  SD before chemoradiation | 2
  PD before chemoradiation | 1
  SD before surgery | 2

3. Secondary Outcome: Histopathologic Tumor Response
Description: Estimate the rate of good histopathologic response as the proportion of grade I and II responders. The analysis population for this objective is the ITT population. Any patient for whom a surgical sample is not available will be considered a poor-responder.
Time Frame: at the time of surgery
Population: Only subjects who had surgery were included in this outcome measure.
Measure: Number; unit: grade II responder
Arm/Group | Chemotherapy, Chemoradiation, Surgery
Number analyzed (Participants) | 1
grade II responder | 1

4. Secondary Outcome: Time to Recurrence:
Description: Time to recurrence is defined as the time from surgical resection to disease recurrence or death from any cause. Patients who have not recurred at the end of follow up will have their recurrence time censored at the last date of contact.
Time Frame: 2 years
Population: The study terminated early, prior to the follow up period being completed. Only one subject had surgery and that subject is still alive at the time of study termination, so time to recurrence cannot be estimated.
Arm/Group | Chemotherapy, Chemoradiation, Surgery
Number analyzed (Participants) | 0

5. Secondary Outcome: Overall Survival:
Description: Overall survival is defined as the time from enrollment to death from any cause. Patients still alive at the end of follow up will have their survival time censored at the last date of contact.
Time Frame: 2 years
Population: The study terminated early, prior to the end of the follow up period for all subjects. At the time of study termination, one subject had expired and the time from enrollment to death for that subject is reported below.
Measure: Number; unit: days
Arm/Group | Chemotherapy, Chemoradiation, Surgery
Number analyzed (Participants) | 1
days | 256

6. Other Pre Specified Outcome: Feasibility Objective
Description: The feasibility of treating patients with localized pancreatic head adenocarcinoma with this neoadjuvant regimen will be evaluated by estimating the proportion of patients completing five of six planned doses. The analysis population will be the ITT population.
Time Frame: From enrollment to end of chemotherapy part of the study
Population: The number of subjects who had 5-6 doses of neoadjuvant regimen
Measure: Number; unit: participants
Arm/Group | Chemotherapy, Chemoradiation, Surgery
Number analyzed (Participants) | 3
participants | 3

7. Other Pre Specified Outcome: CTC Analysis
Description: To evaluate and describe CTC numbers, CTC phenotype characteristics and effectiveness/rate of CTC culturing techniques from patients with pancreatic adenocarcinoma.
Time Frame: End of study
Population: The CTC analysis was added as an amendment. No subjects were enrolled to the study after this amendment was approved, so data for this outcome was not collected or analyzed.
Arm/Group | Chemotherapy, Chemoradiation, Surgery
Number analyzed (Participants) | 0

8. Other Pre Specified Outcome: CTC Expression
Description: To determine and evaluate the correlation between expression or biomarkers in the CTCs and expression of biomarkers in resected tissue specimens within the same cancer patient.
Time Frame: 2 years
Population: The CTC expression endpoint was added as an amendment. No subjects were enrolled to the study after this amendment was approved, so data for this outcome was not collected or analyzed.
Arm/Group | Chemotherapy, Chemoradiation, Surgery
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Start of treatment to end of treatment.
Description: AEs are reported from the start of chemotherapy to the end of study treatment. Any medically significant AEs, which are ongoing at the end of study treatment should be followed until the event is resolved or considered stable.
Arm/Group | Chemotherapy, Chemoradiation, Surgery
Serious Adverse Events (participants affected / at risk) | 2/3
Other Adverse Events (participants affected / at risk) | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Chemotherapy, Chemoradiation, Surgery (N=3)
bile duct stenosis (Hepatobiliary disorders) | 1 (1)
abdominal pain (Gastrointestinal disorders) | 1 (1)
chills (General disorders) | 1 (1)
fever (General disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Chemotherapy, Chemoradiation, Surgery (N=3)
anemia (Blood and lymphatic system disorders) | 1 (1)
leukocytosis (Blood and lymphatic system disorders) | 1 (1)
ear infection (Ear and labyrinth disorders) | 1 (1)
diarrhea (Gastrointestinal disorders) | 2 (2)
nausea (Gastrointestinal disorders) | 2 (2)
vomiting (Gastrointestinal disorders) | 2 (2)
fatigue (General disorders) | 3 (3)
chills (General disorders) | 1 (1)
fever (General disorders) | 1 (1)
pain (General disorders) | 2 (2)
non-cardiac chest pain (General disorders) | 1 (1)
ALT increased (Investigations) | 1 (1)
alkaline phosphatase increase (Investigations) | 1 (1)
AST increased (Investigations) | 1 (1)
blood bilirubin increase (Investigations) | 1 (1)
abnormal appetite (Metabolism and nutrition disorders) | 1 (1)
hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1)
hypokalemia (Metabolism and nutrition disorders) | 1 (1)
dizziness (Nervous system disorders) | 1 (1)
syncope (Nervous system disorders) | 1 (1)
anxiety (Psychiatric disorders) | 1 (1)
insomnia (Psychiatric disorders) | 1 (1)
dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1)
ECRP (Surgical and medical procedures) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes